CLINICAL TRIAL: NCT05022823
Title: Decongestive Progressive Resistance Exercise With Advanced Compression for Breast Cancer Related Lymphedema Management (DREAM): A Randomized Control Trial
Brief Title: Exercise and Compression for Lymphedema
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IIT-0016
Record Dates: First submitted 2021-08-16; First posted 2021-08-26 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: Decongestive Progressive Resistance Exercise; compression sleeve during exercise; adjustable compression garment
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (Active Comparator): Group A (Control). Home decongestive exercise regimen + daytime use of a compression sleeve (12 hours per day)
  Interventions: Device: Compression sleeve, daytime wear; Behavioral: Home exercise program
- DPRE + compression sleeve during exercise (Experimental): Group B. Decongestive Progressive Resistance Exercise + compression sleeve use during exercise + daytime use of a compression sleeve (12 hours per day)
  Interventions: Device: Compression sleeve, worn during exercise; Device: Compression sleeve, daytime wear; Behavioral: Decongestive Progressive Resistance Exercise program
- DPRE + AC garment during exercise (Experimental): Group C. Decongestive Progressive Resistance Exercise + Adjustable Compression (AC) garment use during exercise + daytime use of a compression sleeve (12 hours per day).
  Interventions: Device: Adjustable Compression (AC) garment, worn during exercise; Device: Compression sleeve, daytime wear; Behavioral: Decongestive Progressive Resistance Exercise program

INTERVENTIONS:
Device: Compression sleeve, worn during exercise — Participants wear their daytime compression sleeve during the DPRE program.
  Arms: DPRE + compression sleeve during exercise
Device: Adjustable Compression (AC) garment, worn during exercise — Participants wear an Adjustable Compression (AC) garment during the DPRE program. Participants will be fitted for an Adjustable Compression garment and instructed in its application by a physical therapist.
  Arms: DPRE + AC garment during exercise
Device: Compression sleeve, daytime wear — Compression sleeve worn for at least 12 hours per day, seven days a week.
Behavioral: Decongestive Progressive Resistance Exercise program — Supervised DPRE exercise program, twice a week for 12 weeks. Exercises will be individualized and offered in a group-based format.
  After the 12-week intervention, participants will continue the same program (independently) twice weekly for an additional 12 weeks at home or in a community-based fitness center or attend supervised group exercise sessions virtually.
  Other Names: DPRE
  Arms: DPRE + AC garment during exercise; DPRE + compression sleeve during exercise
Behavioral: Home exercise program — Participants are provided with a home exercise program that follows the decongestive exercise sequence and instructed to perform the exercise sequence once daily for a 10-15 minute period.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to investigate the benefit of combining resistance exercise with use of a compression sleeve on arm lymphedema. In the study, participants will be taught a resistance exercise that follows the decongestive exercise sequence. This program is called "decongestive progressive resistance exercise" (DPRE). To evaluate the benefit from use of a compression garment on the arm. Some participants will wear their usual compression sleeve during exercise and others will use an adjustable compression wrap. The investigators hope to see if this type of combined program is helpful for women with lymphedema. The investigators also want to see if there are benefits from the addition of use of an adjustable compression wrap during exercise over use of a regularly prescribed compression sleeve.

ELIGIBILITY:
Inclusion Criteria:

1. Is a female with a history of breast cancer;
2. Has undergone surgery, including sentinel lymph node biopsy or axillary lymph node dissection;
3. Has visible and palpable unilateral mild to moderate BCRL of at least 200 ml inter-limb volume difference (full limb) or regional lymphedema: defined as a minimal volume difference of 100 ml or 5% in a segment of the arm (e.g. hand and forearm region, elbow and upper arm) after correcting for arm dominance;
4. Has chronic lymphedema, defined as lymphedema that has been present for at least 3 months;
5. Is in the lymphedema maintenance phase of conservative treatment;
6. Uses a well fitted compression sleeve (not older than 1 month) and is agreeable to wear the sleeve for a minimum of 12 hours per day (providing a minimum of 30 mm Hg of pressure);
7. Is agreeable to discontinuing other lymphedema treatments that are beyond standard care, including manual lymph drainage and intermittent pneumatic compression during the 12-week RCT period of the study.
8. Is able to read and understand English.

Exclusion Criteria:

1. Are undergoing or are scheduled to receive chemotherapy or radiotherapy
2. Presents with limb infection/ cellulitis, deep vein thrombosis, or have active metastatic disease;
3. Has any neurological or cognitive deficit, is pregnant, uses a pacemaker, or has other uncontrolled health condition that may interfere with assessment and/or the progressive resistance exercise training intervention;
4. Has any contraindications related to wearing compression on the limb, including arterial insufficiency or congestive heart failure;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Change in Lymphedema Arm Volume | Up to 24 weeks
  Lymphedema will be objectively measured using the optoelectronic limb volumeter (perometer).

SECONDARY OUTCOMES:
Change in Extracellular Fluid Volume | Up to 24 weeks
  Bioimpedance analysis (BIA) is specially designed to estimate extracellular fluid volume in the limb. BIA measures the impedance ratio of the affected and unaffected limb and the resulting calculated index provides an estimate of extracellular fluid volume.
Change in Muscle Strength | Up to 24 weeks
  Muscle strength will be assessed with the one-repetition maximum (1-RM) method for bench press, leg press, and seated row. The 1-RM is the highest weight that can be lifted once using proper form, a smooth motion and without pain or other symptoms.
Change in Grip Strength | Up to 24 weeks
  The Jamar hydraulic hand dynamometer will be used to measure grip strength.
Change in Shoulder Range of Motion | Up to 24 weeks
  Shoulder range of motion (ROM) will be measured using plastic goniometer and each arm will be measured separately for flexion, abduction, internal, external rotation, and horizontal abduction.
Health-Related Quality of Life (Lymph-ICF) | Up to 24 weeks
  The Lymphedema Functioning, Disability, and Health (Lymph-ICF) questionnaire consists of 29 questions related to functional impairments, activity limitations, and participation restrictions in patients with upper limb lymphedema.The total score of the Lymph-ICF on the five areas ranges from 0 to 100, with a score of 0 meaning no impact and higher scores indicative of worse function or negative impact.
Health-Related Quality of Life (SF-36) | Up to 24 weeks
  The Rand Short Form-36 Version 2 (SF-36) questionnaire is comprised of 36 questions that aim to evaluate the following eight models of HRQOL: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality/energy, social functioning, role limitations due to emotional problems, and general mental health.
Physical Activity Level | Up to 24 weeks
  The Godin leisure-time exercise questionnaire (GLTEQ) will be used to assess the physical activity level. The Godin questionnaire is a self reported measure of the average duration and frequency of strenuous (heart beats rapidly), moderate (not exhausting), and mild activities (minimal effort), resistance training, and flexibility training exercise.
Exercise and Compression Adherence | Up to 24 weeks
  Participants will be asked to record their adherence to their assigned exercise and compression intervention program using a daily diary.The adherence diary will collect details on exercise sessions performed each day, including sets, repetitions, and resistance weight, as well as use of the assigned compression sleeve (i.e. use of the garment during exercises and number of hours per day and days per week the compression sleeve is worn).

CONTACTS AND LOCATIONS:
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Al Onazi MM, Campbell KL, Thompson RB, Ghosh S, Mackey JR, Muir A, McNeely ML. Decongestive progressive resistance exercise with an adjustable compression wrap for breast cancer-related lymphoedema (DREAM): protocol for a randomised controlled trial. BMJ Open. 2022 Apr 4;12(4):e053165. doi: 10.1136/bmjopen-2021-053165. PMID 35379618
- See also: Link to the pilot study — https://www.clinicaltrials.gov/ct2/show/NCT02992782?term=NCT02992782&draw=2&rank=1